CLINICAL TRIAL: NCT04320979
Title: Postmastectomy Prophylactic Internal Mammary Nodal Irradiation for High-risk Patients With Non-metastatic Breast Cancer
Brief Title: Postmastecomy Internal Mammary Nodal Irradiation for High-risk Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Shanghai Zhongshan Hospital (Other); Zhejiang Cancer Hospital (Other); Beijing Hospital (Other Government); Liaoning Cancer Hospital & Institute (Other); Jilin Provincial Tumor Hospital (Other); Tangshan People's Hospital (Other); The First Hospital of Jilin University (Other); West China Hospital (Other); Peking Union Medical College Hospital (Other); Henan Cancer Hospital (Other Government); Zhongnan Hospital (Other); Peking University Cancer Hospital & Institute (Other); Fudan University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Air Force Military Medical University, China (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Lanzhou University First Hospital (Unknown); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Principal Investigator, Shulian Wang, Clinical professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/317-2101
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast neoplasm; mastectomy; radiotherapy; internal mammary node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal mammary nodal irradiation (Experimental): chest wall/whole breast and supraclavicular nodal+-axillary plus internal mammary nodal irradiation
  Interventions: Radiation: internal mammary nodal irradiation
- no-internal mammary nodal irradiation (Active Comparator): ipsilateral chest wall/whole breast and supraclavicular +-axillary nodal irradiation
  Interventions: Radiation: no internal mammary nodal irradiation

INTERVENTIONS:
Radiation: internal mammary nodal irradiation — chest wall/whole breast and supraclavicular +-axillary plus internal mammary nodal irradiation (50 Gy in 25 fractions or 43.5Gy in 15 fractions). Patients treated with breast-conserving surgery will receive tumor bed boost. Concurrent boost (60 Gy in 25 fractions over 5 weeks or 49.5 Gy in 15 fractions over 3 weeks) or sequential boost (10 Gy in 5 fractions over 1 week or 8.7 Gy in 3 fractions over 3 days) is optional.
  Arms: internal mammary nodal irradiation
Radiation: no internal mammary nodal irradiation — chest wall/whole breast and supraclavicular+-axillary nodal irradiation (50 Gy in 25 fractions or 43.5Gy in 15 fractions). Concurrent boost (60 Gy in 25 fractions over 5 weeks or 49.5 Gy in 15 fractions over 3 weeks) or sequential boost (10 Gy in 5 fractions over 1 week or 8.7 Gy in 3 fractions over 3 days) is optional.
  Arms: no-internal mammary nodal irradiation

SUMMARY:
The purpose of this study is to evaluate the impact of internal mammary nodal irradiation on disease-free survival in high-risk breast cancer patients treated with mastectomy or breast-conserving surgery.

DETAILED DESCRIPTION:
Eligible patients are randomized into 2 groups: chest wall/whole breast and supraclavicular nodal +-axillary plus internal mammary nodal irradiation, and chest wall/whole breast and supraclavicular nodal +-axillary nodal irradiation. The prescription dose is 50 Gy in 25 fractions over 5 weeks or 43.5Gy in 15 fractions over 3 weeks. Breast cancer patients treated with breast-conserving surgery will receive tumor bed boost.

During and after radiotherapy, the patients are followed and the efficacy and toxicities of radiotherapy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status Scale 0-2
* Histologically confirmed invasive breast cancer
* Underwent total mastectomy/breast-conserving surgery and axillary dissection(10 or more axillary lymph nodes detected) and negative margins
* Patients who had ≥4 positive axillary lymph nodes; or 1-3positive axillary lymph nodes and T3-4; or 1-3positive axillary lymph nodes and T1-2, and score≥3 based on the following high risk factors: age≤40 years(score 1), primary tumor in the inner quadrant (score 1), 2-3 positive axillary lymph nodes (score 1), positive vascular invasion (score 1), re-staged based on eighth Cancer Staging System staging system(IB-IIA score 1， IIB-IIIA score 2); or ypN+ after neoadjuvant chemotherapy
* No supraclavicular or internal mammary nodes metastases based on images before system therapy
* No distant metastases
* Could tolerate radiotherapy
* Treated with chemotherapy (anthracycline and/or taxane-based combined chemotherapy, ≥6 cycles)
* Anticipated to receive endocrine therapy for 5 years if indicated
* Anticipated to receive anti-HER2 therapy for 1 years if indicated
* LVEF≥50% based on echocardiogram
* Willing to follow up
* Written,informed consent

Exclusion Criteria:

* Simultaneous bilateral breast cancer
* Sentinel lymph node biopsy only without axillary dissection
* Had received internal mammary node dissection
* No imaging assessment of the internal mammary nodal before system therapy
* One-stage breast reconstruction
* Severe cardiac insufficiency; myocardial infarction or uncorrected unstable arrhythmia or uncorrected unstable angina in the last 3 months; pericardial disease
* Had history of chest wall or supraclavicular radiotherapy
* Had simultaneous or previous secondary malignancies, except for non-malignant melanoma skin cancer, papillary thyroid / follicular carcinoma, cervical carcinoma in situ, contralateral non-invasive breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years
  failure: relapse of ipsilateral chest wall/breast, axilla, supraclavicular and internal mammary nodal or distant metastasis or contralateral invasive breast cancer or death due to any cause.

SECONDARY OUTCOMES:
overall survival | 5 years
  the incidence of death due to any cause.
cumulative internal mammary nodal recurrence | 5 years
  ipsilateral internal mammary nodal relapse during follow up.
cumulative locoregional recurrence | 5 years
  ipsilateral chest wall/breast, axilla, supraclavicular and internal mammary nodal relapse during follow up.
distant metastasis | 5 years
  the incidence of first relapse beyond locoregional region.
contralateral non-invasive breast cancer or other malignant tumors | 5 years
  the incidence of contralateral invasive breast cancer or other malignant tumors developed after enrollment.
major cardiovascular events | 5 years
  the incidence of death due to coronary heart disease or other heart disease, development of myocardial infarction, coronary recanalization, or hospitalization for a major cardiovascular events (such as heart failure, valvular disease, arrhythmia, unstable angina, or other major cardiovascular event).
incidence of adverse events | 5 years
  graded according to radiation therapy oncology group (RTOG) radiation injury criteria and National Cancer Institute CTCAE version 3.0.
quality of life | 5 years
  questionaire analysis with European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and QLQ-BR23 scale

OTHER OUTCOMES:
Exploratory Translational Research | 5 year
  Circulating blood markers in relation to efficacy and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Shu-lian Wang, M.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Ye-xiong Li, M.D, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Owing to concerns regarding patient privacy.

REFERENCES:
- [Derived] Zhao XR, Fang H, Tang Y, Hu ZH, Jing H, Liang L, Yan XN, Song YW, Jin J, Liu YP, Chen B, Tang Y, Qi SN, Li N, Lu NN, Men K, Hu C, Zhang YH, Li YX, Wang SL. POstmastectomy radioThErapy in Node-posiTive breast cancer with or without Internal mAmmary nodaL irradiation (POTENTIAL): a study protocol for a multicenter prospective phase III randomized controlled trial. BMC Cancer. 2021 Nov 6;21(1):1185. doi: 10.1186/s12885-021-08852-y. PMID 34742270